CLINICAL TRIAL: NCT05975411
Title: Telemedicine Anesthesia Consultation, Pilot Study in Obstetrics.
Acronym: CATmedO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 18-180
Record Dates: First submitted 2023-07-25; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Pregnancy Related
MeSH Terms: interventions — Telemedicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- telemedecine cabin: Anesthesia Consultation with telemedicine cabin installed in Dozulé
  Interventions: Other: Anesthesia Consultation with telemedicine
- telemedicine trolley: Anesthesia Consultation with telemedicine by way of the telemedicine trolley installed in a center close to their place of residence
  Interventions: Other: Anesthesia Consultation with telemedicine
- standard: Anesthesia Consultation at the CHU de Caen as usual.

INTERVENTIONS:
Other: Anesthesia Consultation with telemedicine — Anesthesia Consultation with telemedicine
  Groups: telemedecine cabin; telemedicine trolley

SUMMARY:
Pilot study in Lower Normandy concerning a total of 90 patients scheduled for a pre-anaesthesia consultation in obstetrics. These parturients who plan to give birth at the maternity hospital of the CHU will be invited to carry out their anesthesia consultation with a view to childbirth either by way of the telemedicine cabin installed in Dozulé, or by way of the telemedicine trolley installed in a center close to their place of residence, or at the CHU de Caen as usual.

The validation of the adequacy of the possibilities of telemedicine with the requirements of the anesthesia consultation worked upstream is the main objective of this work, the appreciation of the parturient at this consultation, the appreciation of the consulting and validating professionals will also be collected with the aim of a maximum optimization of this new offer intended for the region.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman
* over 18 years old
* beneficiary of social security/CMU
* Non-emergency pre-anesthesia consultation
* delivery planned at the maternity ward of the University Hospital of Caen
* living in the vicinity of Dozulé or living near an establishment with a telemedicine cart equipped with the necessary equipment
* Having received clear and honest information about the study, and having given their consent
* Having given their consent for a telemedicine consultation
* patient without comorbidity

Exclusion Criteria:

* Patient refusal
* Patient under guardianship
* Patient with psychomotor disability; hearing impaired; visually impaired
* Difficulties in understanding information, expression; foreign language
* Pathological pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnancy
Study Population: pregnancy women
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
assessment of the airways via a telemedicine device | baseline
  * Composite score (rated from 5 to 14) evaluating the risk of difficult orotracheal intubation which is based on the five main elements of the airway evaluation during the anesthesia consultation which are:
  * Mouth opening
  * Mallampati score
  * Cervical spine mobility
  * Thyro-chin distance
  * Patient Profile
  * Lip test

CONTACTS AND LOCATIONS:
Locations (1):
- CAEN University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No